CLINICAL TRIAL: NCT02837809
Title: Early Lung Cancer Detection With Spiral Computed Tomography (CT), Positron Emission Tomography (PET) and Biomarkers: Randomized Trial in High Risk Individuals
Brief Title: Early Lung Cancer Detection in High Risk Individuals
Acronym: MILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT 53/05
Record Dates: First submitted 2016-07-01; First posted 2016-07-20 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: low-dose computed tomography; lung; randomized controlled trial; neoplasms; screening; smoking
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Low Dose CT, annual or biennial, associated with primary prevention and pulmonary function test evaluation.
  Interventions: Radiation: Low dose CT
- Control (No Intervention): Program of primary prevention with pulmonary function test evaluation

INTERVENTIONS:
Radiation: Low dose CT — annual CT vs biennial CT
  Other Names: LDCT
  Arms: Intervention

SUMMARY:
The MILD project is a randomized lung cancer screening trial whose primary aim is to evaluate the impact on mortality of early lung cancer detection through LDCT (low-dose computed tomography) in 2 groups: a control group undergoing a program of primary prevention with pulmonary function test evaluation and a group undergoing a periodic spiral CT associated with primary prevention and pulmonary function test evaluation. This last one is also randomized in two arms: yearly low-dose CT vs CT every 2 years.

MILD trial comprehensive design combines for the first time primary prevention (smoking cessation) with early detection, and molecular risk profile through assessing the value of blood and tissue biomarkers.

DETAILED DESCRIPTION:
The preliminary results of the pilot study on early lung cancer detection by spiral CT and PET launched in Milan in 2000 and published in the Lancet in 2003 showed a positive outcome, confirming the essential safety of spiral CT and a high proportion (95%) of complete resections and stage I disease (77%). However, the results at six years revealed a different picture, with an increasing number of advanced lung cancers being detected from the third to the fifth year, and no evidence of significant mortality reduction for lung cancer by annual CT monitoring of our cohort of heavy smokers. These data were confirmed by a meta-analysis conducted by two senior epidemiologists of Memorial Sloan-Kettering Cancer Center, Peter Bach and Colin Begg, of the three concurrent single arms studies: IEO/INT, Mayo Clinic and Lee Moffitt Cancer Center trials. Such a meta-analysis demonstrated that annual CT increases by 3-4 fold the number of detected lung cancers but does not reduce the incidence of advanced and potentially lethal disease. These data strengthen the validity of the plan to continue clinical research on early lung cancer detection by a randomized controlled study in 2005. In fact there is an overwhelming consensus in the International scientific community that uncontrolled observational studies will not be able to provide further knowledge in this field. Only large randomised controlled clinical trial will hopefully provide convincing evidence on the magnitude of the benefit achievable by early detection programmes with spiral CT in heavy smokers.

In 2005, with the support of AIRC (Italian Association for Cancer Research) and the Ministry of Health, the investigators launched the new INT (National Institute of Tumors) randomized controlled study, named Multicentric Italian Lung Detection trial (MILD), combining smoking cessation with early diagnosis and biologic assessment of individual risk of lung cancer.

The initial goal at INT was to recruit 10,000 subjects from 10 different Italian centres by the end of 2008. This task has proven unfeasible for a number of reasons, including the lack of available institutions with sufficient experience and logistic facilities to run large long-term trials, and the strong campaign in the media in favor of early detection programmes, which has made the randomisation in a control arm unacceptable for a large proportion of volunteers. As a matter of fact, despite the formal collaboration of Istituto Superiore di Sanità (ISS Rome), signed in February 2006, and the acceptance of the protocol by the Ethics Committee of many Italian centres, only two other Institutions have started active accrual by July 2007.

As a consequence, the INT has decided to increase its target for the MILD trial to 4000 subjects, with the aim of joining the other two Italian randomized studies (DANTE and ITALUNG) to provide a strong Italian meta-analysis of at least 10,000 subjects, that might in the future be compared with the two large on-going randomised trials, the NCI trial in the United States and the Nelson trial in northern Europe (Netherlands, Belgium, Denmark), providing concurrent data on the southern European population.

MILD study recruits subjects randomized in 2 groups: a control group undergoes to a program of primary prevention with pulmonary function test evaluation and a group to periodic spiral CT associated with primary prevention and pulmonary function test evaluation. The last one is randomized in two arms: yearly low-dose CT vs CT every 2 years. MILD trial comprehensive design combines for the first time primary prevention with early detection and molecular risk profiling representing an innovative research against lung cancer.

The investigators recruited volunteers through a newspaper and television campaign, that provided information about the study design and eligibility criteria. The participants were asked to sign written informed consent to randomization in one of the two groups. Upon arrival, subjects were given a questionnaire to be completed and returned before leaving the centre. It includes a brief personal and family medical history, smoking details and information about attempts and assistance to stop smoking. A blood sample is collected from each subject at baseline and every two years follow-up. A basic spirometry is performed on each occasion.

Randomization:

* Control group protocol Control group undergo a program of primary prevention with pulmonary function test evaluation and blood collection. Each participant is contacted annually to collect relevant data on health status, hospital admission, and diagnosis or treatment of any concurrent disease, with particular emphasis on respiratory disorders and interval cancers. The study database is updated in real time with all such information.
* CT scan group protocol Baseline and annual single-slice spiral CT are performed without contrast material, with a low-dose protocol, and reconstruction with lung algorithm at every 1 and 5 mm. The CT scanner is a 16 slice. Effective radiation dose is equivalent to 1.54 mSv (milliSievert). Examinations are independently reported by two radiologists within 6 days, on a dedicated workstation and standard lung and mediastinum windows and maximum projection visual resolution reconstruction, for between-observer variability testing. A sophisticate algorithm for volumetric reconstruction and CAD (Computer-Aided Detection) software are used. Investigators deem calcified nodules or lesions with a maximum diameter of 5 mm (measured on lung window) non-suspicious and schedule repeat low-dose CT at next year, as per the protocol. Spiral thin-section CT limited to the area of interest and further examinations for growth assessment are completed within 3 months of baseline CT in every case of non-calcified lesion larger than 5 mm. Non-calcified lesions of 7 mm or larger, are tested with fluorine-18-labelled fluorodeoxyglucose PET(positron emission tomography) and calculation of standardised uptake value. For each patient, the metabolic activity of the lung nodule is assessed by standardised uptake values, measured with regions of interest manually drawn around the nodule on transaxial images.

Blood sample and plasma collection In both groups a sample of peripheral blood is collected during the first evaluation. Five aliquots of 1 millilitre of whole blood are frozen at -80°C.

The aim of biomarker and proteomic analysis and evaluation of individual genetic lung cancer risk is to assess whether this analysis can identify individuals at higher risk of cancer, improve the sensitivity and specificity of imaging techniques, such as low-dose CT scan and PET scan, or both. A team of research nurses, a data manager, and the study coordinator have maintained continuous contact with the enrolled volunteers to guarantee an appropriate follow-up. Each participant is recalled at least twice yearly to collect relevant data on health status, hospital admission, and diagnosis or treatment of any concurrent disease, with particular emphasis on respiratory disorders and interval cancers. The study database is updated in real time with all such information.

In both groups, pulmonary function tests is evaluated with a spirometer connected to a computer for the analysis of data. The following parameters are registered: forced vital capacity (FVC), forced expiratory volume (FEV), the amount of air you exhale may be measured at 1 second (FEV1), forced expiratory flow 25% to 75%, peak expiratory flow (PEF).

People who have even a brief counselling session with a health care professional are more likely to quit smoking. The ASK, ADVISE, ASSESS, ASSIST, and ARRANGE model was developed to help health care professionals with their patients who smoke. The physician asks the patient about their smoking status at every visit; advises the patient to stop smoking; assesses the patient's willingness to quit; assists the patient by setting a date to quit smoking, provides self-help materials, and recommends use of nicotine replacement therapy (such as the nicotine patch); and arranges for follow-up visits.

At present, blood sample aliquots have been collected and stored in the MILD tissue bank, as well as the cancer and healthy tissue samples from all surgically resected cases.

Also the strong commitment to biological research is been boosted by increasing the spectrum of MILD-related studies, covering proteomic and micro-arrays analysis, and launching a new research initiative aimed at evaluation of the role of COPD (Chronic obstructive pulmonary disease) in lung cancer development, with particular interest to the structural, morphologic and proteomic inflammatory damages related to lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smokers, age ≥50 years or older with a minimum of 20 pack-years smoking history, no history of malignant disease, and adequate performance status (assessed on the basis of the patient's eligibility to undergo thoracic surgery).

Exclusion Criteria:

* History of malignant disease in the previous years and not adequate performance status (assessed on the basis of the patient's eligibility to undergo thoracic surgery).

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4099 (Actual)
Dates: Start 2005-09; Primary Completion 2011-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Lung cancer mortality | 10 years
  evaluate the impact on mortality of early lung cancer detection through LDCT at annual or biennial intervals versus no screening

SECONDARY OUTCOMES:
Smoking cessation | 10 years
  evaluate the impact on smoking cessation of early lung cancer detection through LDCT at annual or biennial intervals versus no screening
Molecular risk profile through assessing the value of circulating DNA in blood samples | 10 years
  Circulating DNA, quantified through a real-time quantitative PCR approach based on the 5' nucleotide method: Correlation of results of qPCR DNA levels, epidemiological data on smoking exposition and level of functional impairment (spirometry and DLCO) to define a map of individual biological damage and define a quantitative score of individual risk of lung cancer, possibly related to preneoplastic lung lesions.
Molecular risk profile through assessing the value of microRNA in blood and tissue samples | 10 years
  MicroRNA expression profile, using TaqMan microfluidic cards: Association with aggressiveness of the disease and poor survival in tumors and in normal lung tissue and the critical influence of a smoking related lung microenvironment on tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Pastorino, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sozzi G, Roz L, Conte D, Mariani L, Andriani F, Lo Vullo S, Verri C, Pastorino U. Plasma DNA quantification in lung cancer computed tomography screening: five-year results of a prospective study. Am J Respir Crit Care Med. 2009 Jan 1;179(1):69-74. doi: 10.1164/rccm.200807-1068OC. Epub 2008 Sep 11. PMID 18787214
- [Background] Sozzi G, Pastorino U, Croce CM. MicroRNAs and lung cancer: from markers to targets. Cell Cycle. 2011 Jul 1;10(13):2045-6. doi: 10.4161/cc.10.13.15712. No abstract available. PMID 21623159
- [Background] Boeri M, Pastorino U, Sozzi G. Role of microRNAs in lung cancer: microRNA signatures in cancer prognosis. Cancer J. 2012 May-Jun;18(3):268-74. doi: 10.1097/PPO.0b013e318258b743. PMID 22647364
- [Result] Marchiano A, Calabro E, Civelli E, Di Tolla G, Frigerio LF, Morosi C, Tafaro F, Ferri E, Sverzellati N, Camerini T, Mariani L, Lo Vullo S, Pastorino U. Pulmonary nodules: volume repeatability at multidetector CT lung cancer screening. Radiology. 2009 Jun;251(3):919-25. doi: 10.1148/radiol.2513081313. Epub 2009 Apr 20. PMID 19380692
- [Result] Roz L, Verri C, Conte D, Miceli R, Mariani L, Calabro' E, Andriani F, Pastorino U, Sozzi G. Plasma DNA levels in spiral CT-detected and clinically detected lung cancer patients: a validation analysis. Lung Cancer. 2009 Nov;66(2):270-1. doi: 10.1016/j.lungcan.2009.08.011. Epub 2009 Sep 9. No abstract available. PMID 19744743
- [Result] Sverzellati N, Ingegnoli A, Calabro E, Randi G, La Vecchia C, Marchiano A, Kuhnigk JM, Hansell DM, Zompatori M, Pastorino U. Bronchial diverticula in smokers on thin-section CT. Eur Radiol. 2010 Jan;20(1):88-94. doi: 10.1007/s00330-009-1515-2. Epub 2009 Jul 14. PMID 19597819
- [Result] Boeri M, Verri C, Conte D, Roz L, Modena P, Facchinetti F, Calabro E, Croce CM, Pastorino U, Sozzi G. MicroRNA signatures in tissues and plasma predict development and prognosis of computed tomography detected lung cancer. Proc Natl Acad Sci U S A. 2011 Mar 1;108(9):3713-8. doi: 10.1073/pnas.1100048108. Epub 2011 Feb 7. PMID 21300873
- [Result] Pastorino U, Rossi M, Rosato V, Marchiano A, Sverzellati N, Morosi C, Fabbri A, Galeone C, Negri E, Sozzi G, Pelosi G, La Vecchia C. Annual or biennial CT screening versus observation in heavy smokers: 5-year results of the MILD trial. Eur J Cancer Prev. 2012 May;21(3):308-15. doi: 10.1097/CEJ.0b013e328351e1b6. PMID 22465911
- [Result] Pastorino U. Current status of lung cancer screening. Thorac Surg Clin. 2013 May;23(2):129-40. doi: 10.1016/j.thorsurg.2013.01.018. PMID 23566965
- [Result] Field JK, van Klaveren R, Pedersen JH, Pastorino U, Paci E, Becker N, Infante M, Oudkerk M, de Koning HJ; European Randomized Screening Trial Group. European randomized lung cancer screening trials: Post NLST. J Surg Oncol. 2013 Oct;108(5):280-6. doi: 10.1002/jso.23383. Epub 2013 Jul 25. PMID 23893464
- [Result] Pastorino U, Sverzellati N. Lung cancer: CT screening for lung cancer--do we have an answer? Nat Rev Clin Oncol. 2013 Dec;10(12):672-3. doi: 10.1038/nrclinonc.2013.198. Epub 2013 Nov 5. No abstract available. PMID 24189470
- [Result] Fortunato O, Boeri M, Verri C, Conte D, Mensah M, Suatoni P, Pastorino U, Sozzi G. Assessment of circulating microRNAs in plasma of lung cancer patients. Molecules. 2014 Mar 10;19(3):3038-54. doi: 10.3390/molecules19033038. PMID 24619302
- [Result] Sozzi G, Boeri M, Rossi M, Verri C, Suatoni P, Bravi F, Roz L, Conte D, Grassi M, Sverzellati N, Marchiano A, Negri E, La Vecchia C, Pastorino U. Clinical utility of a plasma-based miRNA signature classifier within computed tomography lung cancer screening: a correlative MILD trial study. J Clin Oncol. 2014 Mar 10;32(8):768-73. doi: 10.1200/JCO.2013.50.4357. Epub 2014 Jan 13. PMID 24419137
- [Result] Boeri M, Sestini S, Fortunato O, Verri C, Suatoni P, Pastorino U, Sozzi G. Recent advances of microRNA-based molecular diagnostics to reduce false-positive lung cancer imaging. Expert Rev Mol Diagn. 2015 Jun;15(6):801-13. doi: 10.1586/14737159.2015.1041377. Epub 2015 Apr 30. PMID 25924864
- [Result] Hu J, Boeri M, Sozzi G, Liu D, Marchiano A, Roz L, Pelosi G, Gatter K, Pastorino U, Pezzella F. Gene Signatures Stratify Computed Tomography Screening Detected Lung Cancer in High-Risk Populations. EBioMedicine. 2015 Jul 8;2(8):831-40. doi: 10.1016/j.ebiom.2015.07.001. eCollection 2015 Aug. PMID 26425689
- [Result] Sestini S, Boeri M, Marchiano A, Pelosi G, Galeone C, Verri C, Suatoni P, Sverzellati N, La Vecchia C, Sozzi G, Pastorino U. Circulating microRNA signature as liquid-biopsy to monitor lung cancer in low-dose computed tomography screening. Oncotarget. 2015 Oct 20;6(32):32868-77. doi: 10.18632/oncotarget.5210. PMID 26451608
- [Result] Silva M, Galeone C, Sverzellati N, Marchiano A, Calareso G, Sestini S, La Vecchia C, Sozzi G, Pelosi G, Pastorino U. Screening with Low-Dose Computed Tomography Does Not Improve Survival of Small Cell Lung Cancer. J Thorac Oncol. 2016 Feb;11(2):187-93. doi: 10.1016/j.jtho.2015.10.014. Epub 2015 Dec 23. PMID 26845115
- [Result] Pastorino U, Boffi R, Marchiano A, Sestini S, Munarini E, Calareso G, Boeri M, Pelosi G, Sozzi G, Silva M, Sverzellati N, Galeone C, La Vecchia C, Ghirardi A, Corrao G. Stopping Smoking Reduces Mortality in Low-Dose Computed Tomography Screening Participants. J Thorac Oncol. 2016 May;11(5):693-699. doi: 10.1016/j.jtho.2016.02.011. Epub 2016 Feb 24. PMID 26921675
- [Result] Sestini S, Boeri M, Marchiano A, Silva M, Calareso G, Galeone C, Sozzi G, Pastorino U. [Lung cancer screening in high-risk subjects: early detection with LDCT and risk stratification using miRNA-based blood test]. Epidemiol Prev. 2016 Jan-Feb;40(1 Suppl 1):42-50. doi: 10.19191/EP16.1S1.P042.029. Italian. PMID 26951732
- [Result] Infante M, Sestini S, Galeone C, Marchiano A, Lutman FR, Angeli E, Calareso G, Pelosi G, Sozzi G, Silva M, Sverzellati N, Cavuto S, La Vecchia C, Santoro A, Alloisio M, Pastorino U. Lung cancer screening with low-dose spiral computed tomography: evidence from a pooled analysis of two Italian randomized trials. Eur J Cancer Prev. 2017 Jul;26(4):324-329. doi: 10.1097/CEJ.0000000000000264. PMID 27222939
- [Derived] Venkadesh KV, Aleef TA, Scholten ET, Saghir Z, Silva M, Sverzellati N, Pastorino U, van Ginneken B, Prokop M, Jacobs C. Prior CT Improves Deep Learning for Malignancy Risk Estimation of Screening-detected Pulmonary Nodules. Radiology. 2023 Aug;308(2):e223308. doi: 10.1148/radiol.223308. PMID 37526548
- [Derived] Pastorino U, Silva M, Sestini S, Sabia F, Boeri M, Cantarutti A, Sverzellati N, Sozzi G, Corrao G, Marchiano A. Prolonged lung cancer screening reduced 10-year mortality in the MILD trial: new confirmation of lung cancer screening efficacy. Ann Oncol. 2019 Jul 1;30(7):1162-1169. doi: 10.1093/annonc/mdz117. PMID 30937431
- [Derived] Silva M, Sverzellati N, Colombi D, Milanese G, La Vecchia C, Galeone C, Marchiano A, Pastorino U. Pleural plaques in lung cancer screening by low-dose computed tomography: prevalence, association with lung cancer and mortality. BMC Pulm Med. 2017 Nov 25;17(1):155. doi: 10.1186/s12890-017-0506-3. PMID 29178853